CLINICAL TRIAL: NCT00004933
Title: A Phase III Study of Interferon-Refractory Patients With BCR/ABL(+) Chronic Myelogenous Leukemia (CML) Treated With Homoharringtonine (NSC #141633) vs. Hydroxyurea
Brief Title: Homoharringtonine Compared With Hydroxyurea for Chronic Myelogenous Leukemia That Has Not Responded to Interferon Alfa
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Poor accrual
Sponsor: Alliance for Clinical Trials in Oncology (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CALGB-19807; U10CA031946 (NIH); CDR0000067617 (Registry Identifier: NCI Physician Data Query)
Record Dates: First submitted 2000-03-07; First posted 2004-04-28 (Estimated); Last update posted 2016-07-04 (Estimated); Status verified 2016-07

CONDITIONS: Leukemia
Keywords: relapsing chronic myelogenous leukemia; chronic phase chronic myelogenous leukemia; Philadelphia chromosome positive chronic myelogenous leukemia
MeSH Terms: conditions — Leukemia; Leukemia, Myeloid, Chronic-Phase; Leukemia, Myelogenous, Chronic, BCR-ABL Positive | interventions — Hydroxyurea; Homoharringtonine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Homoharringtonine (Experimental)
  Interventions: Drug: Homoharringtonine
- Hydroxyurea (Active Comparator)
  Interventions: Drug: hydroxyurea

INTERVENTIONS:
Drug: hydroxyurea — 0.5 to 5 grams PO per day
  Arms: Hydroxyurea
Drug: Homoharringtonine — 2.5 mg/ sq m/ day CIVI for 14 days
  Arms: Homoharringtonine

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop cancer cells from dividing so they stop growing or die. It is not yet known if homoharringtonine is more effective than hydroxyurea for chronic myelogenous leukemia that has not responded to interferon alfa.

PURPOSE: Randomized phase III trial to compare the effectiveness of homoharringtonine with that of hydroxyurea in treating patients who have chronic myelogenous leukemia that has not responded to interferon alfa.

DETAILED DESCRIPTION:
OBJECTIVES: I. Compare the overall survival of interferon alfa refractory chronic myelogenous leukemia patients treated with homoharringtonine to those treated with hydroxyurea. II. Compare the time to progression of these patients treated with these two drugs. III. Estimate the complete and major cytogenetic response and describe the serial cytogenetics of these patients treated with these two drugs.

OUTLINE: This is a randomized study. Patients are randomized to receive one of two treatments. Arm I: Induction: Patients receive homoharringtonine IV continuously over 24 hours daily for 14 days. Induction continues every 28 days for a maximum of 6 courses or until hematopoietic recovery. Maintenance: Patients receive homoharringtonine IV continuously over 24 hours daily for 5 days. Treatment repeats every 28 days. Arm II: Induction: Patients receive oral hydroxyurea daily for 28 days until acceptable blood counts are achieved. Maintenance: Patients receive oral hydroxyurea daily every 28 days to maintain acceptable blood counts. Treatment in both arms continues for a minimum of 6 courses in the absence of disease progression or unacceptable toxicity. Patients are followed every 6 months for a maximum of 10 years.

PROJECTED ACCRUAL: A total of 480 patients (240 per arm) will be accrued for this study within 4 years.

ELIGIBILITY:
1. Documentation of Disease:

   1.1 Diagnosis of Chronic Myelogenous Leukemia (CML) in chronic phase. Patients in either accelerated or blastic phases are not eligible. Clonal cytogenetic evolution alone does not exclude patients. See Appendix I for definitions of accelerated and blastic phases of CML.

   1.2 Patients in whom a Philadelphia chromosome [t(9;22)] is not detectable by cytogenetic studies are eligible if they meet one of the following criteria:
   * BCR/ABL protein detectable by immunoblotting
   * BCR/ABL rearrangement detectable by Southern blot analysis
   * Polymerase chain reaction (PCR) positive fusion transcripts for BCR/ABL
   * BCR/ABL translocation present by fluorescence in situ hybridization (FISH).
2. Prior Treatment:

   2.1 No previous therapy with homoharringtonine (HHT)

   2.2 No more than six months cumulative (<180 days) of prior hydroxyurea (HU) therapy. However, patients may not have received more than 60 days of HU treatment after failing interferon. Patients with previous intolerance or failure to respond to HU are not eligible.

   2.3 Patients must have failed an adequate trial (5M units/m2/day) of alpha-Interferon (IFN) or IFN/ara-C to be eligible, as defined below (any ONE of the following):
   * Failure to achieve a complete hematologic response after 6 months of IFN therapy.
   * Failure to achieve any cytogenetic response (i.e., still 100% Ph+) after 12 months of IFN therapy.
   * Intolerable adverse effects of IFN therapy after at least one month of IFN treatment. Significant documented toxicity of ≥ grade 3 (using NCI Common Toxicity Criteria guidelines) due to IFN is required.
   * Loss of a prior hematologic remission or cytogenetic response to IFN.
   * A two-fold increase in WBC count when compared to WBC count when IFN therapy was initiated.
3. Age ≥ 16 years
4. Patients with uncontrolled tachyarrhythmias (such as, atrial fibrillation, paroxysmal supraventricular tachycardia, and ventricular tachycardias not adequately controlled) are not eligible.
5. Non-pregnant and non-nursing. Treatment under this protocol would expose an unborn child to significant risks. Women and men of reproductive potential should agree to use an effective means of birth control.

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2000-01; Primary Completion 2001-05 (Actual); Study Completion 2001-05 (Actual)

PRIMARY OUTCOMES:
Overall survival | 4 years

CONTACTS AND LOCATIONS:
Overall Officials: Dan DeAngelo, MD, Study Chair — Dana-Farber Cancer Institute
Locations (133):
- United States (133):
  - Veterans Affairs Medical Center - Birmingham, Birmingham, Alabama
  - MBCCOP - University of South Alabama, Mobile, Alabama
  - CCOP - Greater Phoenix, Phoenix, Arizona
  - Veterans Affairs Medical Center - Phoenix (Hayden), Phoenix, Arizona
  - Veterans Affairs Medical Center - Tucson, Tucson, Arizona
  - Arizona Cancer Center, Tucson, Arizona
  - University of Arkansas for Medical Sciences, Little Rock, Arkansas
  - Veterans Affairs Medical Center - Little Rock (McClellan), Little Rock, Arkansas
  - University of California San Diego Cancer Center, La Jolla, California
  - Veterans Affairs Medical Center - Long Beach, Long Beach, California
  - USC/Norris Comprehensive Cancer Center, Los Angeles, California
  - Jonsson Comprehensive Cancer Center, UCLA, Los Angeles, California
  - Beckman Research Institute, City of Hope, Los Angeles, California
  - Veterans Affairs Outpatient Clinic - Martinez, Martinez, California
  - CCOP - Bay Area Tumor Institute, Oakland, California
  - Chao Family Comprehensive Cancer Center, Orange, California
  - University of California Davis Medical Center, Sacramento, California
  - UCSF Cancer Center and Cancer Research Institute, San Francisco, California
  - Veterans Affairs Medical Center - San Francisco, San Francisco, California
  - CCOP - Santa Rosa Memorial Hospital, Santa Rosa, California
  - David Grant Medical Center, Travis Air Force Base, California
  - Veterans Affairs Medical Center - Denver, Denver, Colorado
  - University of Colorado Cancer Center, Denver, Colorado
  - CCOP - Christiana Care Health Services, Wilmington, Delaware
  - Lombardi Cancer Center, Georgetown University, Washington D.C., District of Columbia
  - Walter Reed Army Medical Center, Washington D.C., District of Columbia
  - CCOP - Mount Sinai Medical Center, Miami Beach, Florida
  - CCOP - Atlanta Regional, Atlanta, Georgia
  - Dwight David Eisenhower Army Medical Center, Fort Gordon, Georgia
  - Cancer Research Center of Hawaii, Honolulu, Hawaii
  - University of Illinois at Chicago Health Sciences Center, Chicago, Illinois
  - Veterans Affairs Medical Center - Chicago (Westside Hospital), Chicago, Illinois
  - University of Chicago Cancer Research Center, Chicago, Illinois
  - CCOP - Central Illinois, Decatur, Illinois
  - Veterans Affairs Medical Center - Hines (Hines Junior VA Hospital), Hines, Illinois
  - Loyola University Medical Center, Maywood, Illinois
  - University of Iowa Hospitals and Clinics, Iowa City, Iowa
  - University of Kansas Medical Center, Kansas City, Kansas
  - CCOP - Wichita, Wichita, Kansas
  - Veterans Affairs Medical Center - Wichita, Wichita, Kansas
  - Veterans Affairs Medical Center - Lexington, Lexington, Kentucky
  - Albert B. Chandler Medical Center, University of Kentucky, Lexington, Kentucky
  - MBCCOP - LSU Medical Center, New Orleans, Louisiana
  - Tulane University School of Medicine, New Orleans, Louisiana
  - Veterans Affairs Medical Center - New Orleans, New Orleans, Louisiana
  - Louisiana State University Health Sciences Center - Shreveport, Shreveport, Louisiana
  - Veterans Affairs Medical Center - Shreveport, Shreveport, Louisiana
  - Veterans Affairs Medical Center - Togus, Togus, Maine
  - Marlene & Stewart Greenebaum Cancer Center, University of Maryland, Baltimore, Maryland
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - Boston Medical Center, Boston, Massachusetts
  - Veterans Affairs Medical Center - Boston (Jamaica Plain), Jamaica Plain, Massachusetts
  - University of Massachusetts Memorial Medical Center, Worcester, Massachusetts
  - Veterans Affairs Medical Center - Ann Arbor, Ann Arbor, Michigan
  - University of Michigan Comprehensive Cancer Center, Ann Arbor, Michigan
  - Veterans Affairs Medical Center - Detroit, Detroit, Michigan
  - Barbara Ann Karmanos Cancer Institute, Detroit, Michigan
  - Henry Ford Hospital, Detroit, Michigan
  - CCOP - Grand Rapids Clinical Oncology Program, Grand Rapids, Michigan
  - Providence Hospital - Southfield, Southfield, Michigan
  - Veterans Affairs Medical Center - Minneapolis, Minneapolis, Minnesota
  - University of Minnesota Cancer Center, Minneapolis, Minnesota
  - Veterans Affairs Medical Center - Biloxi, Biloxi, Mississippi
  - University of Mississippi Medical Center, Jackson, Mississippi
  - Veterans Affairs Medical Center - Jackson, Jackson, Mississippi
  - Keesler Medical Center - Keesler AFB, Keesler Air Force Base, Mississippi
  - Veterans Affairs Medical Center - Columbia (Truman Memorial), Columbia, Missouri
  - Ellis Fischel Cancer Center - Columbia, Columbia, Missouri
  - Veterans Affairs Medical Center - Kansas City, Kansas City, Missouri
  - CCOP - Kansas City, Kansas City, Missouri
  - CCOP - Cancer Research for the Ozarks, Springfield, Missouri
  - St. Louis University Health Sciences Center, St Louis, Missouri
  - Barnes-Jewish Hospital, St Louis, Missouri
  - CCOP - St. Louis-Cape Girardeau, St Louis, Missouri
  - CCOP - Montana Cancer Consortium, Billings, Montana
  - University of Nebraska Medical Center, Omaha, Nebraska
  - CCOP - Southern Nevada Cancer Research Foundation, Las Vegas, Nevada
  - Norris Cotton Cancer Center, Lebanon, New Hampshire
  - Veterans Affairs Medical Center - Albuquerque, Albuquerque, New Mexico
  - MBCCOP - University of New Mexico HSC, Albuquerque, New Mexico
  - Veterans Affairs Medical Center - Buffalo, Buffalo, New York
  - Roswell Park Cancer Institute, Buffalo, New York
  - CCOP - North Shore University Hospital, Manhasset, New York
  - North Shore University Hospital, Manhasset, New York
  - Memorial Sloan-Kettering Cancer Center, New York, New York
  - New York Presbyterian Hospital - Cornell Campus, New York, New York
  - Mount Sinai Medical Center, NY, New York, New York
  - Herbert Irving Comprehensive Cancer Center, New York, New York
  - State University of New York - Upstate Medical University, Syracuse, New York
  - Veterans Affairs Medical Center - Syracuse, Syracuse, New York
  - CCOP - Syracuse Hematology-Oncology Associates of Central New York, P.C., Syracuse, New York
  - Lineberger Comprehensive Cancer Center, UNC, Chapel Hill, North Carolina
  - Veterans Affairs Medical Center - Durham, Durham, North Carolina
  - Duke Comprehensive Cancer Center, Durham, North Carolina
  - CCOP - Southeast Cancer Control Consortium, Winston-Salem, North Carolina
  - Comprehensive Cancer Center of Wake Forest University Baptist Medical Center, Winston-Salem, North Carolina
  - Barrett Cancer Center, The University Hospital, Cincinnati, Ohio
  - Veterans Affairs Medical Center - Cincinnati, Cincinnati, Ohio
  - Cleveland Clinic Taussig Cancer Center, Cleveland, Ohio
  - CCOP - Columbus, Columbus, Ohio
  - Arthur G. James Cancer Hospital - Ohio State University, Columbus, Ohio
  - Veterans Affairs Medical Center - Dayton, Dayton, Ohio
  - CCOP - Dayton, Kettering, Ohio
  - Oklahoma Medical Research Foundation, Oklahoma City, Oklahoma
  - Veterans Affairs Medical Center - Oklahoma City, Oklahoma City, Oklahoma
  - Oregon Cancer Center at Oregon Health Sciences University, Portland, Oregon
  - Veterans Affairs Medical Center - Portland, Portland, Oregon
  - CCOP - Columbia River Program, Portland, Oregon
  - Rhode Island Hospital, Providence, Rhode Island
  - Medical University of South Carolina, Charleston, South Carolina
  - CCOP - Greenville, Greenville, South Carolina
  - CCOP - Upstate Carolina, Spartanburg, South Carolina
  - University of Tennessee, Memphis Cancer Center, Memphis, Tennessee
  - Veterans Affairs Medical Center - Memphis, Memphis, Tennessee
  - Simmons Cancer Center - Dallas, Dallas, Texas
  - Brooke Army Medical Center, Fort Sam Houston, Texas
  - University of Texas Medical Branch, Galveston, Texas
  - Texas Tech University Health Science Center, Lubbock, Texas
  - University of Texas Health Science Center at San Antonio, San Antonio, Texas
  - Veterans Affairs Medical Center - San Antonio (Murphy), San Antonio, Texas
  - Veterans Affairs Medical Center - Temple, Temple, Texas
  - CCOP - Scott and White Hospital, Temple, Texas
  - Huntsman Cancer Institute, Salt Lake City, Utah
  - Veterans Affairs Medical Center - Salt Lake City, Salt Lake City, Utah
  - CCOP - Southwestern Vermont Regional Cancer Center, Bennington, Vermont
  - Vermont Cancer Center, Burlington, Vermont
  - Veterans Affairs Medical Center - White River Junction, White River Junction, Vermont
  - Veterans Affairs Medical Center - Richmond, Richmond, Virginia
  - MBCCOP - Massey Cancer Center, Richmond, Virginia
  - CCOP - Virginia Mason Research Center, Seattle, Washington
  - Swedish Cancer Institute, Seattle, Washington
  - Veterans Affairs Medical Center - Seattle, Seattle, Washington
  - CCOP - Northwest, Tacoma, Washington